CLINICAL TRIAL: NCT03222141
Title: Edwards SAPIEN 3 Transcatheter Heart Valve Therapy for High Risk and Inoperable Patients
Brief Title: PARTNER II Trial: Placement of AoRTic TraNscathetER Valves II - High Risk and Nested Registry 7
Acronym: PII S3HR/NR7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12 S3HR/NR7
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2018-08-14 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: SAPIEN 3; Transfemoral; Transapical; Transaortic; TAVI; Aortic Stenosis; THV; Aortic Valve; Transcatheter Heart Valve; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SAPIEN 3™ valve (Experimental)
  Interventions: Device: TAVR Implantation of the THV Prosthesis

INTERVENTIONS:
Device: TAVR Implantation of the THV Prosthesis — Patients with TAVR implantation
  Other Names: SAPIEN 3™valve

SUMMARY:
The purpose of this trial is to determine the safety and effectiveness of the Edwards SAPIEN 3 transcatheter heart valve and delivery systems which are intended for use in patients with symptomatic, calcific, severe aortic stenosis, and are in high risk.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center trial for patients undergoing aortic valve replacement with the Edwards SAPIEN 3 THV for severe aortic stenosis. Patient cohorts will include those inoperable and those considered as a high surgical risk (STS ≥8%). The study also includes NR7 patients (patients with a 20mm vessel size).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s and an initial aortic valve area (AVA) of ≤0.8 cm2 or indexed EOA < 0.5 cm2/m2. Qualifying echo must be within 60 days of the date of the procedure.
2. Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
3. The heart team agrees (and verified in the case review process) that valve implantation will likely benefit the patient.
4. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
5. The study patient agrees to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which will be conducted as a phone follow-up.
6. STS > 8

Exclusion Criteria:

1. Pre-existing mechanical or bioprosthetic valve in any position.
2. Active bacterial endocarditis within 6 months (180 days) of procedure.
3. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
4. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure. Implantation of a permanent pacemaker or ICD is not considered exclusion criteria.
5. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University
Locations (40):
- United States (39):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center DC, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Indiana University Health-Methodist Hospital, Indianapolis, Indiana
  - The University of Iowa, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence St.Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Austin Heart, PLLC, Austin, Texas
  - Medical City Dallas, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
- St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vincent F, Thourani VH, Ternacle J, Redfors B, Cohen DJ, Hahn RT, Li D, Crowley A, Webb JG, Mack MJ, Kapadia S, Russo M, Smith CR, Alu MC, Leon MB, Pibarot P. Time-of-Day and Clinical Outcomes After Surgical or Transcatheter Aortic Valve Replacement: Insights From the PARTNER Trials. Circ Cardiovasc Qual Outcomes. 2022 Jan;15(1):e007948. doi: 10.1161/CIRCOUTCOMES.121.007948. Epub 2022 Jan 18. PMID 35041482
- [Derived] Ong G, Pibarot P, Redfors B, Weissman NJ, Jaber WA, Makkar RR, Lerakis S, Gopal D, Khalique O, Kodali SK, Thourani VH, Anwaruddin S, McAndrew T, Zhang Y, Alu MC, Douglas PS, Hahn RT. Diastolic Function and Clinical Outcomes After Transcatheter Aortic Valve Replacement: PARTNER 2 SAPIEN 3 Registry. J Am Coll Cardiol. 2020 Dec 22;76(25):2940-2951. doi: 10.1016/j.jacc.2020.10.032. PMID 33334422
- [Derived] Chen S, Redfors B, O'Neill BP, Clavel MA, Pibarot P, Elmariah S, Nazif T, Crowley A, Ben-Yehuda O, Finn MT, Alu MC, Vahl TP, Kodali S, Leon MB, Lindman BR. Low and elevated B-type natriuretic peptide levels are associated with increased mortality in patients with preserved ejection fraction undergoing transcatheter aortic valve replacement: an analysis of the PARTNER II trial and registry. Eur Heart J. 2020 Feb 21;41(8):958-969. doi: 10.1093/eurheartj/ehz892. PMID 31883339
- [Derived] Summers MR, Leon MB, Smith CR, Kodali SK, Thourani VH, Herrmann HC, Makkar RR, Pibarot P, Webb JG, Leipsic J, Alu MC, Crowley A, Hahn RT, Kapadia SR, Tuzcu EM, Svensson L, Cremer PC, Jaber WA. Prosthetic Valve Endocarditis After TAVR and SAVR: Insights From the PARTNER Trials. Circulation. 2019 Dec 10;140(24):1984-1994. doi: 10.1161/CIRCULATIONAHA.119.041399. Epub 2019 Nov 6. PMID 31690104

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAPIEN 3™ Valve
Started | 583
Completed (30-day Follow-up) | 565
Not Completed | 18
Not completed — Death | 15
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | SAPIEN 3™ Valve
Number analyzed (Participants) | 583
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245
  Male | 338
STS score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 8.6 (3.7)
NYHA III/IV [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  Participants | 525
Coronary artery disease [Count of Participants; unit: Participants] | 444

OUTCOME MEASURES:

1. Primary Outcome: The Composite Rate of All-cause Mortality, All Stroke, and AI ≥ Moderate
Description: The composite rate of all-cause mortality, all stroke, and AI ≥ moderate for patients deemed as 'high risk' using the Edwards SAPIEN 3 transcatheter heart valve (THV).
Time Frame: 30 Days
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | SAPIEN 3™ Valve
Number analyzed (Participants) | 583
percentage of patients | 6.7 [5.1 to 8.6]

2. Secondary Outcome: Number of Participants With Major Vascular Complications
Description: The rate of major vascular complications at 30 days post implantation
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Groups:
- SAPIEN 3™ THV: TAVR Implantation of the THV Prosthesis: Patients with TAVR implantation
Arm/Group | SAPIEN 3™ THV
Number analyzed (Participants) | 583
Participants | 29

3. Secondary Outcome: Number of Participants With Aortic Insufficiency at 30 Days
Description: The proportion of patients with aortic insufficiency ≥ moderate at 30 days.
Time Frame: 30 Days
Population: Echo data was available only for 532 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3™ Valve
Number analyzed (Participants) | 532
Participants | 16

ADVERSE EVENTS:
Time Frame: the adverse event data was collected over 30 days
Groups:
- SAPIEN 3™ THV: TAVR Implantation of the THV Prosthesis: Patients with TAVR implantation.
  High risk cohort
Arm/Group | SAPIEN 3™ THV
All-Cause Mortality (participants affected / at risk) | 13/583
Serious Adverse Events (participants affected / at risk) | 232/583
Other Adverse Events (participants affected / at risk) | 397/583
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN 3™ THV (N=583)
Any Adverse Event (Investigations) | 6 (7)
Access site and access related vascular injury - Aortic root rupture (Injury, poisoning and procedural complications) | 2 (2)
Access site and access related vascular injury - Dissection (Injury, poisoning and procedural complications) | 5 (5)
Access site and access related vascular injury - Distal embolization (noncerebral) from vascular sou (Injury, poisoning and procedural complications) | 1 (1)
Access site and access related vascular injury - Failure of percutaneous access site closure (Injury, poisoning and procedural complications) | 5 (5) — Resulting in intervention
Access site and access related vascular injury - Hematoma (Injury, poisoning and procedural complications) | 5 (5)
Access site and access related vascular injury - Other (Injury, poisoning and procedural complications) | 2 (2)
Access site and access related vascular injury - Perforation (Injury, poisoning and procedural complications) | 1 (1)
Access site and access related vascular injury - Pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (4)
Access site and access related vascular injury - Stenosis (Injury, poisoning and procedural complications) | 2 (2)
Access site and access related vascular injury - Thoracic aortic dissection (Injury, poisoning and procedural complications) | 1 (1)
Access site and access related vascular injury - Ventricular rupture (Apical rupture) (Injury, poisoning and procedural complications) | 1 (1)
Anemia/Hemolytic anemia (Blood and lymphatic system disorders) | 5 (5)
Angina/Cardiac chest pain (Cardiac disorders) | 1 (1)
Aortic insufficiency/Regurgitation PV leak - Non structural dysfunction (Cardiac disorders) | 5 (5)
Aortic insufficiency/Regurgitation non valvular cause (Cardiac disorders) | 1 (1)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 105 (108)
Bleeding - Hemorrhage (General disorders) | 41 (44)
Cardiac arrest (Cardiac disorders) | 8 (9)
Cardiac tamponade (Cardiac disorders) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1)
Device embolization (Injury, poisoning and procedural complications) | 1 (1)
Device migration/malposition requiring intervention (Injury, poisoning and procedural complications) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Exercise intolerance or weakness (Metabolism and nutrition disorders) | 1 (1)
Gastro Intestinal event - Non-hemorrhagic (Gastrointestinal disorders) | 10 (10)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 2 (2)
Heart failure/CHF/Low output failure (Cardiac disorders) | 29 (31)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
Infection - Access site infection (Infections and infestations) | 1 (1)
Infection - Bacteremia (Infections and infestations) | 2 (2)
Infection - Other (Infections and infestations) | 1 (1)
Infection - Respiratory infection (Infections and infestations) | 7 (7)
Infection - Sepsis (Infections and infestations) | 2 (2)
Infection - Urinary tract infection (Renal and urinary disorders) | 6 (6)
Ischemia (Investigations) | 1 (1)
MI (Cardiac disorders) | 3 (3)
Mental state change (not neurological) - Confusion (Psychiatric disorders) | 3 (3)
Mental state change (not neurological) - Depression (Psychiatric disorders) | 3 (3)
Miscellaneous - Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Miscellaneous - Fall (Injury, poisoning and procedural complications) | 2 (2)
Miscellaneous - Other (General disorders) | 1 (1)
Musculoskeletal - Fracture (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal - Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neurological - Dysphasia/Aphasia (Nervous system disorders) | 1 (1)
Neurological - Hemiparesis (One sided body weakness) (Nervous system disorders) | 1 (1)
Neurological - Ischemic stroke (Nervous system disorders) | 7 (7)
Neurological - Sensory loss on one side of body (Nervous system disorders) | 1 (1)
Neurological - TIA (Nervous system disorders) | 3 (3)
Neurological - Undetermined stroke (Investigations) | 1 (1)
Renal insufficiency or renal failure (Renal and urinary disorders) | 15 (15)
Respiratory event - Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory event - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory event - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory event - Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Respiratory event - Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Syncope (Vascular disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Thromboembolic event (Surgical and medical procedures) | 2 (2)
Unknown cause of death (Investigations) | 1 (1)
Vascular complication - Non-access related (Vascular disorders) | 4 (4)
Other (Investigations) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN 3™ THV (N=583)
Abnormal lab value (Investigations) | 71 (82)
Anemia/Hemolytic anemia (Blood and lymphatic system disorders) | 54 (54)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 128 (146)
Bleeding - Hemorrhage (Vascular disorders) | 118 (126)
Heart failure/CHF/Low output failure (Cardiac disorders) | 41 (41)
Renal insufficiency or renal failure (Renal and urinary disorders) | 54 (54)
Thrombocytopenia (Blood and lymphatic system disorders) | 40 (40)
Other (Investigations) | 41 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No